CLINICAL TRIAL: NCT02995512
Title: Mechanistic Effects of Colchicine in Patients With Myocardial Infarction A Single Center Phase 4 Single Arm Open-label Study Evaluating the FDA-approved Drug, Colchicine, at the FDA-approved Gout Dose in Patients With Myocardial Infarction
Brief Title: Mechanistic Effects of Colchicine in Patients With Myocardial Infarction
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: feasibility
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-01704
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; colchicine; anti-inflammatory
MeSH Terms: conditions — Myocardial Infarction | interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Myocardial Infarction (MI) Patients (Experimental)
  Interventions: Drug: Colchicine 0.6 mg tablets

INTERVENTIONS:
Drug: Colchicine 0.6 mg tablets — 1.2 mg PO followed by 0.6 mg PO 1 hour later

SUMMARY:
The aim of this study is to determine the immuno-modulatory mechanistic effects of colchicine in patients with myocardial infarction (MI). Investigators hypothesize that colchicine exerts its anti-inflammatory properties by switching the metabolism of neutrophils, thereby reducing the expression of adhesion molecules responsible for their recruitment in MI.

DETAILED DESCRIPTION:
This is a pilot study to explore the mechanistic effects of colchicine in patients with MI. The study will be conducted sequentially in 3 parts:

1. Blood will be collected from up to 10 healthy volunteers for protocol development. (Group 1).
2. Blood will be collected from 20 MI patients within 24 hours of presentation at New York University (NYU) Langone Medical Center and Bellevue Hospital Center (BHC). Neutrophil adhesion to human aortic endothelial cells, quantitative expression of adhesion molecules on the surface of neutrophils, quantitative levels of adhesion molecules on neutrophils and endothelial cells, and neutrophil metabolism, using a Seahorse Analyzer will be evaluated pre- and post-addition of in vitro colchicine. (Group 2)
3. The standard low-dose loading regimen of colchicine (1.2 mg followed by 0.6 mg one hour later) will be administered to 20 patients with MI at BHC. Blood will be collected prior to drug administration, 2 to 3 hours after completion of the colchicine load, and 23 to 24 hours after the completion of the colchicine load. Neutrophil adhesion to human aortic endothelial cells, quantitative expression of adhesion molecules on the surface of neutrophils, quantitative levels of adhesion molecules on neutrophils and endothelial cells, and neutrophil metabolism will be evaluated pre- and post-addition of in vitro colchicine (exact markers will be determined based on the results of in viro studies above). (Group 3)

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age for the healthy volunteer subset.
* 18 years of age and within 24 hours of an MI for the MI subset.

Exclusion Criteria:

Subjects in all 3 groups will be excluded if they meet one of the following criteria

* history of myelodysplasia;
* Use of anti-inflammatory medications, with the exception of aspirin, within 5 half-lives;
* medications known to interact with colchicine;
* known creatinine clearance <30 cc/minute (severe kidney disease);
* pregnant; or
* Unable to consent.

MI subjects who will have oral colchicine administered will have the following additional exclusion criteria:

* history of intolerance to colchicine;
* acute or chronic symptoms of diarrhea within 72 hours prior to enrollment;
* hemoglobin <10 g/dL or clinical evidence of active bleeding during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
Number of neutrophils adherent to TNFα-stimulated endothelial cells | 1 Day
  Metabolism of neutrophils will be measured using the Seahorse assay.

SECONDARY OUTCOMES:
Levels of adhesion molecules on neutrophils and endothelial cells quantified using PCR | 1 Day
  Metabolism of neutrophils will be measured using the Seahorse assay.
Expression of adhesion molecules on the surface of neutrophils assessed via flow cytometry | 1 Day
  Measurements of L-selectin, CD11b, and active CD11b will be made via an Accuri C6 flow cytometer using standard antibodies on an aliquot of whole blood.
Measures of neutrophil metabolism (e.g. O2 consumption) | 1 Day
  Metabolism of neutrophils will be measured using the Seahorse assay.

CONTACTS AND LOCATIONS:
Overall Officials: Binita Shah, MD, Principal Investigator — NYU Langone Health